CLINICAL TRIAL: NCT01086267
Title: A Phase 1/2 Study of BMS-908662 (XL281) Alone or in Combination With Cetuximab in Subjects With K-RAS or B-RAF Mutation Positive Advanced or Metastatic Colorectal Cancer
Brief Title: Safety and Efficacy Study of BMS-908662 Alone or in Combination With Cetuximab in Subjects With K-RAS or B-RAF Mutation Positive Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA206-001; 2010-018944-15 (EudraCT Number)
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — BMS 908662; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- BMS-908662 (A1) (Experimental): Phase 1
  Interventions: Drug: BMS-908662
- Cetuximab (A1) (Experimental): Phase 1
  Interventions: Drug: Cetuximab
- BMS-908662 (B1) (Experimental): Phase 2
  Interventions: Drug: BMS-908662
- BMS-908662 + Cetuximab (B2) (Experimental): Phase 2
  Interventions: Drug: BMS-908662; Drug: Cetuximab

INTERVENTIONS:
Drug: BMS-908662 — Capsules, Oral, escalating doses starting at 25 mg, every 12 hours (Q 12 h), Continuously
  Arms: BMS-908662 (A1)
Drug: BMS-908662 — Capsules, Oral, (TBD) mg, Q 12 h, Continuously
  Arms: BMS-908662 (B1); BMS-908662 + Cetuximab (B2)
Drug: Cetuximab — Vial, IV, 400 mg/m² loading dose followed by 250 mg/m² maintenance dose, Weekly, Continuously
  Arms: BMS-908662 + Cetuximab (B2); Cetuximab (A1)

SUMMARY:
The purpose of the study is to identify a safe and tolerable dose of BMS-908662 in combination with cetuximab; and then to evaluate the tumor response to BMS-908662 when administered alone or in combination with cetuximab

DETAILED DESCRIPTION:
Phase 1: Single Arm Study

Phase 2: Randomized Controlled, Parallel

ELIGIBILITY:
Inclusion Criteria:

* Subjects with K-RAS (codon 12 or 13) or B -RAF (V600E) mutation positive advanced or metastatic colorectal cancer who have relapsed or are refractory to 2 or more standard systemic anticancer regimes for metastatic disease, or are intolerant to existing therapies.
* Histologic or cytologic confirmation of the diagnosis.
* Eastern Cooperative Oncology Group (ECOG) ≤ 1
* Adequate organ & marrow function.

Exclusion Criteria:

* Uncontrolled or significant cardiovascular disease.
* Phase 2: Prior therapy with a RAF inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Toxicity will be evaluated according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 3 | Assessments every 1-2 weeks while receiving study drug

SECONDARY OUTCOMES:
Efficacy as determined by estimates of objective response rates and response duration | Efficacy measured at least every 8 weeks while receiving study drug
Pharmacodynamics (PD) will be assessed by evaluating markers of RAS/RAF pathway activity | PD assessed during the first 4 weeks on study
Pharmacokinetics (PK) for BMS-908662 as determined by minimum observed concentrations [Cmin]. | PK measured during first 4 weeks on study
Pharmacokinetics (PK) for BMS-908662 as determined by maximum observed concentrations [Cmax]. | PK measured during first 4 weeks on study
Pharmacokinetics (PK) for BMS-908662 as determined by time of maximum observed concentration [Tmax]. | PK measured during first 4 weeks on study
Pharmacokinetics (PK) for BMS-908662 as determined by area under the concentration-curve for one dosing interval [AUC(TAU)]. | PK measured during first 4 weeks on study
Pharmacokinetics (PK) for BMS-908662 as determined by accumulation index [AI]. | PK measured during first 4 weeks on study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (2):
  - Oncology Research Associates D/B/A, Scottsdale, Arizona
  - Usc Norris Comprehensive Cancer Center, Los Angeles, California
- Local Institution, Ottawa, Ontario, Canada

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx